CLINICAL TRIAL: NCT02973204
Title: Circulating Tumor Cells and Tumor DNA in HCC and NET - Patient-specific Biomarkers for Clinical Decision Support and Tailored Relapse Diagnostics
Brief Title: Circulating Tumor Cells and Tumor DNA in HCC and NET
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SK-HCC-NET
Record Dates: First submitted 2016-11-18; First posted 2016-11-25 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular; Neuroendocrine Tumors
Keywords: tumor DNA; circulating tumor cells; biopsy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neuroendocrine Tumors; Neoplastic Cells, Circulating | interventions — Sorafenib; Radiofrequency Ablation; Everolimus; lanreotide; Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples and biopsies when available.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HCC sorafenib: HCC patients referred for Sorafenib treatment
  Interventions: Drug: Sorafenib
- HCC curative treatment: HCC patient undergoing potential curative treatment, eg. radiofrequency ablation (RFA) or resection
  Interventions: Procedure: Radiofrequency ablation (RFA) or surgery
- NET everolimus: Pancreatic NET patients referred for Everolimus treatment
  Interventions: Drug: Everolimus
- NET ssta: Small intestinal or unknown primary NET patients referred for treatment with somatostatin analogues, eg. lanreotide and octreotide
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Sorafenib
  Other Names: Nexavar; Anatomical Therapeutic Chemical Classification System L01XE05
  Groups: HCC sorafenib
Procedure: Radiofrequency ablation (RFA) or surgery — Intended curative surgery or RFA
  Groups: HCC curative treatment
Drug: Everolimus
  Other Names: Certican; Afinitor; Votubia; Anatomical Therapeutic Chemical Classification System L01XE10
  Groups: NET everolimus
Drug: Lanreotide — Or other somatostatin analogues (SSTA), eg. Sandostatin
  Other Names: Ipstyl; Sandostatin LAR; Octreotide
  Groups: NET ssta

SUMMARY:
Background Treatment and control of cancer is associated with high costs, to patients in the form of side effects and discomfort during investigations, to society in the form of expensive drugs and studies.

Circulating tumor cells (CTC) has received great attention as a cancer biomarker in trying to estimate future course in patients with breast cancer, colon cancer and prostate cancer. CTC is believed to be a crucial step in cancer spreading to the bloodstream and giving rise to metastases. Detection of circulating tumor DNA (ctDNA) specifically adds specificity to the analysis of the CTC.

The investigators would like to with molecular biological methods predict which patients requires special monitoring and individualized therapy and explore these tests as clinical decision support.

Purpose and method

In a blood sample from patients with neuro-endocrine tumor (NET) and hepatocellular carcinoma (HCC), the investigators will by cell separation, flow cytometry and DNA sequencing and digital polymerase chain reaction (PCR):

1. Identify and isolate the CTC and investigate these for tumor-specific mutations.
2. Quantify ctDNA and analyze this for specific mutations, which in the past has been found frequent in NET and HCC.
3. Compare findings of mutations on CTC and ctDNA with mutations in tissue biopsies.

The results are compared with the clinical data on disease course, including the effect of treatment and survival.

Subjects 40 Patients with small intestinal/unknown primary NET before treatment with somatostatin analogues 30 patients with pancreatic NET before treatment with Everolimus 30 patients with presumed radically treated HCC 30 patients with HCC in treatment with Sorafenib A blood sample will be taken prior to the start of treatment, after 1 month after start of treatment and thereafter every 3.-6. month for up to two years.

Perspectives In several cancer types molecular diagnostics have had significant influence in treatment and control strategy. The goal is in future to be able to take advantage of a so-called "liquid biopsy" as clinical decision support. The study will bring new knowledge to this growing field of research.

ELIGIBILITY:
Inclusion Criteria:

* one of the above mentioned diseases
* planed surgery, RFA, Somatostatin Analogue, Sorafenib or Everolimus treatment
* signed informed consent

Exclusion Criteria:

* age below 18, concomitant invasive cancer (not skin cancer) and planed emigration of Denmark.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 patients newly diagnosed NET patients referred for somatostatin analogue treatment for small intestinal NET or NET with unknown primary.
  30 Pancreatic NET patients treated for known residual disease will be monitored for possible progression of disease and response to Everolimus 30 HCC patients supposed radically treated, either by RFA or liver resection, will be followed with regard to relapse.
  30 HCC patients treated with Sorafenib monitored for treatment response
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2016-11; Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Concordance between specific DNA mutations found in patient biopsies and plasma circulating tumor DNA | 2 months
  Methods: digital droplet PCR and targeted sequencing of blood samples and biopsies

SECONDARY OUTCOMES:
Flow cytometry for detection and quantification of CTC in peripheral blood (absolute and relative counts) | 3 years
Correlations between mutations found in circulating tumor DNA and amount of circulating tumor cells and treatment response according to RECIST criteria | up to 5 years
  Methods: digital droplet PCR and targeted sequencing of blood samples, and flowcytometry and cell separation of blood samples
Correlations between mutations found in circulating tumor DNA and amount of circulating tumor cells and survival | up to 5 years
  Methods: digital droplet PCR and targeted sequencing of blood samples, and flowcytometry and cell separation of blood samples
Correlations between mutations fund in circulating DNA and circulating tumor cells | 3 years
  Methods: digital droplet PCR and targeted sequencing of blood samples, and flowcytometry and cell separation of blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kelsen, Consultant, Study Chair — Department of Hepatology and Gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology and Gastroenterology, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janson ET, Sorbye H, Welin S, Federspiel B, Gronbaek H, Hellman P, Ladekarl M, Langer SW, Mortensen J, Schalin-Jantti C, Sundin A, Sundlov A, Thiis-Evensen E, Knigge U. Nordic guidelines 2014 for diagnosis and treatment of gastroenteropancreatic neuroendocrine neoplasms. Acta Oncol. 2014 Oct;53(10):1284-97. doi: 10.3109/0284186X.2014.941999. Epub 2014 Aug 20. PMID 25140861
- [Background] Bruix J, Sherman M; American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma: an update. Hepatology. 2011 Mar;53(3):1020-2. doi: 10.1002/hep.24199. No abstract available. PMID 21374666
- [Background] Zhang Y, Li J, Cao L, Xu W, Yin Z. Circulating tumor cells in hepatocellular carcinoma: detection techniques, clinical implications, and future perspectives. Semin Oncol. 2012 Aug;39(4):449-60. doi: 10.1053/j.seminoncol.2012.05.012. PMID 22846862
- [Background] Khan MS, Tsigani T, Rashid M, Rabouhans JS, Yu D, Luong TV, Caplin M, Meyer T. Circulating tumor cells and EpCAM expression in neuroendocrine tumors. Clin Cancer Res. 2011 Jan 15;17(2):337-45. doi: 10.1158/1078-0432.CCR-10-1776. Epub 2011 Jan 11. PMID 21224371
- [Background] Khan MS, Kirkwood A, Tsigani T, Garcia-Hernandez J, Hartley JA, Caplin ME, Meyer T. Circulating tumor cells as prognostic markers in neuroendocrine tumors. J Clin Oncol. 2013 Jan 20;31(3):365-72. doi: 10.1200/JCO.2012.44.2905. Epub 2012 Dec 17. PMID 23248251
- [Background] Schulze K, Gasch C, Staufer K, Nashan B, Lohse AW, Pantel K, Riethdorf S, Wege H. Presence of EpCAM-positive circulating tumor cells as biomarker for systemic disease strongly correlates to survival in patients with hepatocellular carcinoma. Int J Cancer. 2013 Nov;133(9):2165-71. doi: 10.1002/ijc.28230. Epub 2013 Jun 11. PMID 23616258
- [Background] Guo W, Yang XR, Sun YF, Shen MN, Ma XL, Wu J, Zhang CY, Zhou Y, Xu Y, Hu B, Zhang X, Zhou J, Fan J. Clinical significance of EpCAM mRNA-positive circulating tumor cells in hepatocellular carcinoma by an optimized negative enrichment and qRT-PCR-based platform. Clin Cancer Res. 2014 Sep 15;20(18):4794-805. doi: 10.1158/1078-0432.CCR-14-0251. Epub 2014 Jul 9. PMID 25009297
- [Background] Francis JM, Kiezun A, Ramos AH, Serra S, Pedamallu CS, Qian ZR, Banck MS, Kanwar R, Kulkarni AA, Karpathakis A, Manzo V, Contractor T, Philips J, Nickerson E, Pho N, Hooshmand SM, Brais LK, Lawrence MS, Pugh T, McKenna A, Sivachenko A, Cibulskis K, Carter SL, Ojesina AI, Freeman S, Jones RT, Voet D, Saksena G, Auclair D, Onofrio R, Shefler E, Sougnez C, Grimsby J, Green L, Lennon N, Meyer T, Caplin M, Chung DC, Beutler AS, Ogino S, Thirlwell C, Shivdasani R, Asa SL, Harris CR, Getz G, Kulke M, Meyerson M. Somatic mutation of CDKN1B in small intestine neuroendocrine tumors. Nat Genet. 2013 Dec;45(12):1483-6. doi: 10.1038/ng.2821. Epub 2013 Nov 3. PMID 24185511
- [Background] Jiao Y, Shi C, Edil BH, de Wilde RF, Klimstra DS, Maitra A, Schulick RD, Tang LH, Wolfgang CL, Choti MA, Velculescu VE, Diaz LA Jr, Vogelstein B, Kinzler KW, Hruban RH, Papadopoulos N. DAXX/ATRX, MEN1, and mTOR pathway genes are frequently altered in pancreatic neuroendocrine tumors. Science. 2011 Mar 4;331(6021):1199-203. doi: 10.1126/science.1200609. Epub 2011 Jan 20. PMID 21252315
- [Background] Marinoni I, Kurrer AS, Vassella E, Dettmer M, Rudolph T, Banz V, Hunger F, Pasquinelli S, Speel EJ, Perren A. Loss of DAXX and ATRX are associated with chromosome instability and reduced survival of patients with pancreatic neuroendocrine tumors. Gastroenterology. 2014 Feb;146(2):453-60.e5. doi: 10.1053/j.gastro.2013.10.020. Epub 2013 Oct 19. PMID 24148618
- [Background] Pipinikas CP, Dibra H, Karpathakis A, Feber A, Novelli M, Oukrif D, Fusai G, Valente R, Caplin M, Meyer T, Teschendorff A, Bell C, Morris TJ, Salomoni P, Luong TV, Davidson B, Beck S, Thirlwell C. Epigenetic dysregulation and poorer prognosis in DAXX-deficient pancreatic neuroendocrine tumours. Endocr Relat Cancer. 2015 Jun;22(3):L13-8. doi: 10.1530/ERC-15-0108. Epub 2015 Apr 21. No abstract available. PMID 25900181
- [Background] Rimassa L, Santoro A. Sorafenib therapy in advanced hepatocellular carcinoma: the SHARP trial. Expert Rev Anticancer Ther. 2009 Jun;9(6):739-45. doi: 10.1586/era.09.41. PMID 19496710
- [Background] Schulze K, Imbeaud S, Letouze E, Alexandrov LB, Calderaro J, Rebouissou S, Couchy G, Meiller C, Shinde J, Soysouvanh F, Calatayud AL, Pinyol R, Pelletier L, Balabaud C, Laurent A, Blanc JF, Mazzaferro V, Calvo F, Villanueva A, Nault JC, Bioulac-Sage P, Stratton MR, Llovet JM, Zucman-Rossi J. Exome sequencing of hepatocellular carcinomas identifies new mutational signatures and potential therapeutic targets. Nat Genet. 2015 May;47(5):505-511. doi: 10.1038/ng.3252. Epub 2015 Mar 30. PMID 25822088
- [Background] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- [Background] Sorensen BS, Wu L, Wei W, Tsai J, Weber B, Nexo E, Meldgaard P. Monitoring of epidermal growth factor receptor tyrosine kinase inhibitor-sensitizing and resistance mutations in the plasma DNA of patients with advanced non-small cell lung cancer during treatment with erlotinib. Cancer. 2014 Dec 15;120(24):3896-901. doi: 10.1002/cncr.28964. Epub 2014 Aug 7. PMID 25103305
- [Background] Neychev V, Steinberg SM, Cottle-Delisle C, Merkel R, Nilubol N, Yao J, Meltzer P, Pacak K, Marx S, Kebebew E. Mutation-targeted therapy with sunitinib or everolimus in patients with advanced low-grade or intermediate-grade neuroendocrine tumours of the gastrointestinal tract and pancreas with or without cytoreductive surgery: protocol for a phase II clinical trial. BMJ Open. 2015 May 19;5(5):e008248. doi: 10.1136/bmjopen-2015-008248. PMID 25991462